CLINICAL TRIAL: NCT01488786
Title: A Study to Evaluate the Safety and Efficacy of the BrainPort® Vision Device in Subjects Who Are Blind
Brief Title: A Study to Evaluate the BrainPort® Vision Device in Subjects Who Are Blind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wicab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: WCB1-010
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Blindness
Keywords: Assistive Technology; Non-Surgical Visual Prosthetic; Sensory Substitution
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BrainPort Vision Device (Experimental): Single Arm
  Interventions: Device: BrainPort Vision Device

INTERVENTIONS:
Device: BrainPort Vision Device — 2-3 days of training (10 hours) followed by minimum in-home use 300 minutes per month for 12 months.

SUMMARY:
The purpose of this study is to assess the safety of the BrainPort vision device and to demonstrate improved object recognition and word identification and ambulation with use of the BrainPort vision device in subjects who are medically documented as blind, with acuity of 20/ 5000 or worse.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed written medical or low vision diagnosis of No Light Perception or Light Perception
* Performance on the FrACT acuity test of worse than 20/5000 or impossible to measure.
* Minimum post 6 months diagnosis blindness.
* Previously completed conventional rehabilitation such as orientation and mobility training with a cane or guide dog.
* Able to have read to him or her, understand, and sign the informed consent form.
* Daily access to an accessible computer with email for study communication, device- use logging and access to device user manual preferred.
* Willing and able to complete all testing, training, and follow- up evaluations required by the study protocol, after receiving a short orientation on the use of the device.

Exclusion Criteria:

* Current oral health problems as determined from the oral health exam which preclude enrollment in the study in the judgment of the Principal Investigator.
* Any medical condition that would interfere with performance on the assessments.
* Prior use of the BrainPort vision device.
* Known neuropathies of tongue or skin tactile system.
* Smoke or chew tobacco products less than 12 months prior to study enrollment
* Any allergies to nickel or stainless steel
* History of seizures or epilepsy.
* If female, pregnant. Women of child bearing potential must agree to use appropriate birth control to prevent pregnancy for the duration of the study.
* People with implanted electrical medical devices (i.e. pacemaker, deep brain stimulator, cochlear implant).
* Psychiatric disease including anxiety disorders and forms of depression (using provided Beck Anxiety Inventory (BAI) and Beck Depression Inventory (BDI- II) as screening tools).
* Any disease or condition that prevents understanding or communication of informed consent, study demands and testing protocols including the following:
* Cognitive decline including forms of dementia and/or progressive neurological disease
* Deafness or selective frequency hearing loss that prevents hearing device alarms and alerts.
* Does not speak English
* Blindness occurring due to cortical injury (i.e. stroke, traumatic brain injury, etc)
* Principal Investigator, in his or her judgment, does not believe the subject is a good candidate for the trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  The primary safety objective is to demonstrate that the rate of clinically significant device-related adverse events is less than 10%. This will require an observed event-free rate of approximately 97%.
Object Recognition | 1 year
  The primary efficacy objective is to demonstrate that at least 50% of subjects achieve a success rate in object recognition exceeding that expected by chance alone.

SECONDARY OUTCOMES:
Word Identification | 1 year
  A secondary efficacy objective is to demonstrate that at least 50% of subjects correctly identify at least 50% of a series of three- to five-letter words.
Ambulation/Mobility | 1 year
  Another secondary efficacy objective is to demonstrate at least 35% of subjects demonstrate sign recognition in a mobility task.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Arnoldussen, Study Director — Wicab, Inc.; William Seiple, Principal Investigator — Lighthouse International
Locations (7):
- United States (6):
  - Independence for the Blind of West Florida Inc., Pensacola, Florida
  - The Chicago Lighthouse for People Who Are Blind and Visually Impaired, Chicago, Illinois
  - Envision, Wichita, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Lighthouse International, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Canadian National Institute for the Blind, Toronto, Canada